CLINICAL TRIAL: NCT06752577
Title: Safety and Tolerability of Vertebral Bone Marrow-derived Mesenchymal Stem Cells (BM-MSC) in Real World Scenarios of Patients With Chronic Kidney Disease (CKD)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Ossium Health, Inc. (Industry)
Responsible Party: Principal Investigator, LaTonya J. Hickson, Division Chair of Nephrology and Hypertension, Mayo Clinic
Other Study IDs: 24-011356
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases; Kidney Transplant
Keywords: stem cells; regenerative medicine; mesenchymal stromal cells; kidney disease; kidney failure; diabetic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Renal Insufficiency; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSC: Individuals with chronic kidney disease (including a kidney transplant that is losing function) will receive allogeneic, bone marrow-derived mesenchymal stem cells (MSC). Two administration routes will be used. Repeat dosing is allowed.
  Interventions: Drug: Allogeneic, vertebral bone marrow-derived mesenchymal stem cells (MSC)

INTERVENTIONS:
Drug: Allogeneic, vertebral bone marrow-derived mesenchymal stem cells (MSC) — 1) intravenous infusion or 2) combined intravenous plus intra-arterial (to kidney) infusion of cells. Total dose: 200x10^6 MSC (administered over 15 minutes to 2 hours). Repeat dosing allowed at 6 month intervals.

SUMMARY:
The purpose of this protocol is to treat an intermediate-sized population with chronic kidney disease (CKD) including kidney transplant recipients. The protocol uses allogeneic bone marrow-derived mesenchymal stem cells (MSCs). MSC infusion may be delivered 1) intravenous or 2) intravenous plus intra-arterial to both kidneys. Individuals will have subsequent follow up for safety evaluations. Repeat dosing is allowed.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2
* Hemoglobin A1c ≤9%, if diabetes mellitus present
* If kidney transplant recipient, must have eGFR<60 mL/min/1.73m2 and evidence of progressive kidney function loss over ≥6 months
* Ability to give informed consent

Exclusion Criteria

* Anemia (hemoglobin <8.5 g/dL)
* Body weight >150 kg or BMI >50
* Uncontrolled hypertension: sustained systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) ≥100 mmHg despite maximal doses of at least 2 different classes of anti-hypertensive medications
* Chronic hypotension history: sustained SBP <85 mmHg
* Kidney failure requiring ongoing kidney replacement therapy including hemodialysis or peritoneal dialysis
* Active, high-dose immunosuppression therapy (e.g. chronic prednisone ≥20 mg daily)
* Solid organ transplantation history; excluding kidney transplant
* Active treatment for acute cellular rejection, in kidney transplant recipients
* Recent cardiovascular event (hospitalization for myocardial infarction, stroke, congestive heart failure (NYHA class ≥III or ejection fraction ≤30%) within 3 months or uncontrolled cardiac arrhythmias (e.g. ventricular arrhythmia, supraventricular tachycardia and bradyarrhythmia)
* History of liver cirrhosis
* Chronic obstructive pulmonary disease or asthma requiring daily medication
* History of recurring blood clotting disorder (thromboembolism: pulmonary embolism, deep venous thrombosis) requiring chronic anticoagulation therapy
* Pregnancy
* Unwilling to use contraception for at least 2 months after MSC infusion if sexually active and able to become pregnant or father a child.
* Active malignancy
* Active infection (e.g. systemic or specific organ involvement such as pneumonia or osteomyelitis; in kidney transplant recipients, active BK nephropathy)
* Recent COVID-19 infection, within the last 1 month
* History of hepatitis B or C (without cure), or HIV infection
* History of allergic reaction to cellular products (i.e. blood transfusions, platelets)
* Active tobacco use
* Illicit drug use and excessive alcohol use
* Presence of psychosocial issues (e.g., uncontrolled mental illness, unpredictable childcare or eldercare responsibilities, irregular/ inflexible work schedule) that may interfere with the ability to complete all study procedures
* Anticipating prolonged travel or other physical restrictions that would prohibit return for scheduled study visits.
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Chronic Kidney Disease (CKD) or Kidney Transplant losing function
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events and/or serious adverse events | 6 months after each MSC infusion
  Number of adverse events and/or serious adverse events associated with mesenchymal stem cell (MSC) intervention

CONTACTS AND LOCATIONS:
Overall Officials: LaTonya J Hickson, MD, Principal Investigator — Nephrology and Hypertension, Mayo Clinic, Jacksonville, Florida
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Hickson LJ, Eirin A, Lerman LO. Challenges and opportunities for stem cell therapy in patients with chronic kidney disease. Kidney Int. 2016 Apr;89(4):767-78. doi: 10.1016/j.kint.2015.11.023. Epub 2016 Jan 26. PMID 26924058
- [Background] Hickson LJ, Herrmann SM, McNicholas BA, Griffin MD. Progress toward the Clinical Application of Mesenchymal Stromal Cells and Other Disease-Modulating Regenerative Therapies: Examples from the Field of Nephrology. Kidney360. 2021 Mar;2(3):542-557. doi: 10.34067/KID.0005692020. PMID 34316720
- [Derived] Patel HA, Wang J, Zinn CJ, Learmonth M, Lerman LO, Wolfram J, Hickson LJ. Fortifying the Diabetic Kidney Disease Treatment Armamentarium: Multitarget Senotherapeutic and Regenerative Strategies. J Am Soc Nephrol. 2025 May 7;36(8):1655-1658. doi: 10.1681/ASN.0000000754. No abstract available. PMID 40333016
- [Derived] Andrews TD, Day GS, Irani SR, Kanekiyo T, Hickson LJ. Uremic Toxins, CKD, and Cognitive Dysfunction. J Am Soc Nephrol. 2025 Jun 1;36(6):1208-1226. doi: 10.1681/ASN.0000000675. Epub 2025 Feb 26. PMID 40009460
- See also: Related Info — https://www.mayo.edu/research/clinical-trials/faculty-search-results?authid=13932080